CLINICAL TRIAL: NCT07196865
Title: Comparison of the Clinical Effects of Open, Closed, and Semi-close Hemorrhoidectomy: Study Protocol for a Single-center, Prospective, Open-label and Randomized Clinical Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHPutianU 2025918
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel-group, randomized controlled trial (RCT). Participants are randomly allocated in a 1:1:1 ratio to one of three distinct intervention groups, where they receive only that specific surgical intervention and are followed concurrently throughout the study period. The groups are defined by the wound management technique used after hemorrhoidectomy:
  Group 1 (Open): Wound left unsutured. Group 2 (Closed):Wound fully closed with interrupted non-absorbable sutures. Group 3 (Semi-Closed): Distal half of the incision closed with interrupted sutures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Hemorrhoidectomy Group (Experimental): Patients in this group will undergo open hemorrhoidectomy. Following external stripping and internal ligation, the wound will be left open without any sutures for healing by secondary intention.
  Interventions: Procedure: Open Hemorrhoidectomy
- Closed Hemorrhoidectomy Group (Experimental): Patients in this group will undergo closed hemorrhoidectomy (Ferguson technique). After achieving hemostasis, the entire wound will be closed primarily using interrupted non-absorbable sutures.
  Interventions: Procedure: Closed Hemorrhoidectomy (Ferguson Technique)
- Semi-Closed Hemorrhoidectomy Group (Experimental): Patients in this group will undergo semi-closed hemorrhoidectomy. Following hemostasis, the distal half of the incision (away from the anal canal) will be closed with interrupted sutures, while the proximal half is left open.
  Interventions: Procedure: Semi-Closed Hemorrhoidectomy

INTERVENTIONS:
Procedure: Open Hemorrhoidectomy — Patients in this group undergo a hemorrhoidectomy procedure where, after external stripping and internal ligation, the surgical wound is left entirely open without sutures to heal by secondary intention. All patients receive standard postoperative care including potassium permanganate rinses and povidone-iodine disinfection.
  Arms: Open Hemorrhoidectomy Group
Procedure: Closed Hemorrhoidectomy (Ferguson Technique) — Patients in this group undergo a hemorrhoidectomy procedure where, after achieving hemostasis, the entire surgical wound is closed primarily using interrupted non-absorbable sutures. All patients receive standard postoperative care including potassium permanganate rinses and povidone-iodine disinfection.
  Arms: Closed Hemorrhoidectomy Group
Procedure: Semi-Closed Hemorrhoidectomy — Patients in this group undergo a hemorrhoidectomy procedure where, after achieving hemostasis, the distal half of the incision (away from the anal canal) is closed with interrupted sutures, while the proximal half remains open. All patients receive standard postoperative care including potassium permanganate rinses and povidone-iodine disinfection.
  Arms: Semi-Closed Hemorrhoidectomy Group

SUMMARY:
This study compares three different ways surgeons close the wound after removing hemorrhoids (piles): leaving it completely open, stitching it completely closed, or stitching only half of it closed (semi-closed). The goal is to see which method leads to faster healing, less pain, fewer complications, and better long-term results. Patients undergoing hemorrhoidectomy will be randomly assigned to one of the three groups. All patients will receive standard post-operative care. Researchers will measure healing time, pain levels, need for pain medication, hospital stay, complications, and check if hemorrhoids come back within one year.

DETAILED DESCRIPTION:
Hemorrhoids are a very common condition, and when surgery is needed, there is no consensus on the best way to manage the surgical wound afterward. This single-center, prospective, randomized clinical trial aims to directly compare the clinical outcomes of the three primary wound management techniques: open, closed, and semi-closed hemorrhoidectomy.

A total of 378 patients will be randomly assigned to one of the three treatment groups. The primary focus is on comparing key short-term outcomes, including the time it takes for the wound to fully heal, the length of the hospital stay, and the rate of complications such as surgical site infection, bleeding, and urinary retention.

Secondary outcomes will provide a broader picture of patient recovery. Pain will be carefully assessed using a standardized pain scale (Visual Analog Scale) on multiple days after surgery and by tracking the total amount of pain medication required during hospitalization. Furthermore, to understand the long-term effectiveness of each technique, the study will follow patients for one year after surgery to assess their quality of life and monitor for any recurrence of hemorrhoids.

This is the first clinical trial to evaluate all three techniques within the same study. The results are expected to provide high-quality evidence to help surgeons choose the most effective wound management strategy, ultimately improving patient care and recovery after hemorrhoid surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years.
2. Clinical diagnosis of mixed hemorrhoids requiring surgical intervention.
3. Scheduled to undergo hemorrhoidectomy with ligation of internal hemorrhoids and excision of external hemorrhoids.
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. History of mental illness or cognitive impairment that may affect the ability to provide informed consent or comply with the study protocol.
2. Diagnosis of diabetes mellitus.
3. Planned concomitant procedures (e.g., radiofrequency ablation, sclerotherapy) in addition to hemorrhoidectomy.
4. Inability or unwillingness to comply with scheduled follow-up visits.
5. Presence of severe perioperative comorbidities that render the patient unsuitable for the planned surgical protocol or anesthesia (as determined by the attending anesthesiologist or surgeon).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | Daily from postoperative Day 1 until complete epithelialization is achieved (assessed for up to 28 days post-surgery)
  The time required for complete wound healing, defined as 100% re-epithelialization of the surgical site with no exudate or scab, assessed by a blinded evaluator.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS score) | Baseline (preoperative), and on postoperative days 1, 2, 3, 5, 7, and 14 (±2 days).
  Pain intensity assessed using the Visual Analog Scale (VAS, 0-10) at rest and during defecation.
Perianal edema severity | Postoperative days 1, 2, 3, 5, 7, and 14 (±2 days).
  Severity of swelling around the surgical site evaluated by trained research nurses using a standardized 0-6 point scale.
Length of hospital stay | From end of surgery until discharge (assessed up to 7 days postoperatively).
  Duration of hospitalization measured in hours from the end of surgery to discharge, using standardized discharge criteria.
Complication incidence | Within 30 days after surgery.
  Occurrence of postoperative complications (e.g., infection, bleeding, urinary retention) classified and graded using the Clavien-Dindo system.